CLINICAL TRIAL: NCT03694873
Title: Oral Tramadol Versus Oral Celecoxib for Post-perineal Repair Analgesia After Spontaneous Vaginal Birth in Obese Women: A Randomised Controlled Trial
Brief Title: Oral Tramadol Versus Oral Celecoxib for Post-perineal Repair Analgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perineal pain
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Perineal Pain
MeSH Terms: interventions — Tramadol; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tramadol (Experimental): one tablet of Tramadol 100 mg (Tramaw, Global Napi, Giza,Egypt) administered orally immediately, 12 h and 24 h after randomization.
  Interventions: Drug: Tramadol Hydrochloride
- celecoxib (Active Comparator): one tablet of Celecoxib 200 mg (Celebrex® 200, Pﬁzer,USA) administered orally immediately, 12 h and 24 h after randomization.
  Interventions: Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: Tramadol Hydrochloride — one tablet of Tramadol 100 mg (Tramaw, Global Napi, Giza,Egypt) administered orally immediately, 12 h and 24 h after randomization.
  Arms: tramadol
Drug: Celecoxib 200mg — Celecoxib 200 mg (Celebrex® 200, Pﬁzer,USA) administered orally immediately, 12 h and 24 h after randomization.
  Arms: celecoxib

SUMMARY:
This trial will be performed to compare the effectiveness of oral tramadol versus oral celecoxib for the management of perineal pain following episiotomy or perineal tear repair after spontaneous vaginal birth in obese women

DETAILED DESCRIPTION:
Pain after episiotomy or tear of perineal tissues during childbirth is often inadequately treated and may be severe. Not only did perineal pain negatively affect the physical and mental functioning of the woman, but also it might decrease the success of breastfeeding and reduced her ability to care for her child. The methods of relieving perineal pain included medication and non-medication. When the perineal pain was mild, the most common analgesic used was acetaminophen. Whereas the perineal pain was more severe, other drugs had been chosen such as opioid, non-opioid, and a combination of both opioid and non-opioid analgesics

ELIGIBILITY:
Inclusion Criteria:

* Age:18-35 years
* Obese women with BMI ≥ 30.
* completed full 37-weeks gestation.
* spontaneous vaginal delivery with medio-lateral episiotomy or perineal tear requiring repair.
* Singleton alive fetus.

Exclusion Criteria:

* known allergy to investigated drugs(tramadol or celecoxib).
* regular use of analgesic drugs before or during pregnancy.
* any medical condition known to be potentially exacerbated by opioids, including alimentary canal disorders, hepatic and renal disease.
* instrumental vaginal delivery.
* 3rd or 4th degree perineal tear.
* severe postpartum haemorrhage (>1,500 ml).
* complicating maternal diseases (pregestational/gestational diabetes mellitus; bleeding disorders; pre-eclampsia and other hypertensive disorders of pregnancy).
* epidural nor combined spinal-epidural analgesia in labour
* a history of peptic ulcer,asthma,thrombocytopaenia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2018-12-05 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
perineal pain | 1 hour after repair of episiotomy
  perineal pain severity using visual analogue scale

SECONDARY OUTCOMES:
perineal pain | 1 hours after repair of episiotomy
  perineal pain severity using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University